CLINICAL TRIAL: NCT01735513
Title: Intraprocedural Intraaortic Embolic Protection With the EmbolX Device in Patients Undergoing Transaortic Transcatheter Aortic Valve Implantation: a Randomized-controlled Trial
Brief Title: Intraprocedural Intraaortic Embolic Protection With the EmbolX Device in Patients Undergoing Transaortic Transcatheter Aortic Valve Implantation
Acronym: TAo-EmbolX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Matthias Thielmann, PD. Dr. med. Matthias Thielmann, West German Heart Center Essen
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: WDHZ-TC-TAo-EmbolX
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Transaortic Transcatheter Aortic Valve Implantation
Keywords: transaortic TAVI or TAVR; embolic protection device; EmbolX; efficacy; during transaortic TAVI; reduce the incidence of new foci of restricted diffusion on diffusion-weighted MRI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transaortic TAVI with EmbolX (Experimental): Subjects are randomized into this arm to receive a transaortic transcatheter aortic valve implantation with the use of the embolic protection device "EmbolX"
  Interventions: Device: Intra-aortic embolic protection management system; Embol-X
- Transaortic TAVI without EmbolX (Active Comparator): Subjects are randomized into this arm to receive a transaortic transcatheter aortic valve implantation without the use of the embolic protection device "EmbolX"
  Interventions: Device: Intra-aortic embolic protection management system; Embol-X

INTERVENTIONS:
Device: Intra-aortic embolic protection management system; Embol-X — The Embol-X system is positioned within the aorta to capture emboli, such as blood clots or tissue fragments, to prevent them from traveling through a patient's bloodstream during TAVI. The EMBOL-X system features a small, expandable, polyester-mesh filtration system that is placed inside the aorta above the aortic clamp during open-heart surgery or transaortic TAVI procedures, where it captures particles in the bloodstream that otherwise might have remained in the patient's circulatory system. A recent presentation characterized the removal of aortic cross-clamps as creating in some patients "embolic showers" which have the potential to cause neurocognitive complications, stroke and other organ damage. In documented procedures, 97% of EMBOL-X system filters showed detectable captured embolic matter, visible proof that the system is removing potentially dangerous emboli from the bloodstream.
  Other Names: Embol-X, Edwards Lifesciences, Irvine, CA, USA. The EMBOL- X intra-aortic embolic management system.

SUMMARY:
Study hypothesis: Reduction of cerebral embolic lesions during transcatheter aortic valve implantation by the use of an embolic protection device.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic severe aortic valve stenosis (valve area <0.8 cm2) are considered candidates for TAVI (TAVR) if they have a logistic European System for Cardiac Operative Risk Evaluation score (EuroSCORE) ≥15% or surgery is deemed to be at excessive risk because of comorbidities and other risk factors not being captured by these scoring systems. Indication for TAVI in the individual patient is discussed in a consensus conference of cardiologists and cardiac surgeons, and patient's or physician's preference alone is not considered adequate for decision making. The performance of TAVI in these patients is approved by the local authorities. All patients have to agree to participate in the study, and written informed consent is obtained.

Exclusion Criteria:

Patients are excluded from TAVI (TAVR) in the presence of any of the following conditions:

* bicuspid aortic valve
* aortic annulus diameter ≤18 or ≥27 mm
* procelain aorta
* unprotected left main disease
* recent myocardial infarction or cerebrovascular event
* sepsis or active endocarditis
* severe aortic atheroma
* left ventricular or atrial thrombus
* active peptic ulcer
* bleeding diathesis
* hypersensitivity to antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The detection of new morphological brain injury with new hyper-intense DW-MRI cerebral lesions on the post-treatment compared to the pretreatment MRI imaging | Postoperative day 1-3
  MRI of the brain is obtained at the same time as clinical exams. Scans are performed on a 1.5-T MR unit and a circular polarized head coil. The imaging protocol includes a transversal DW, single shot echo-planar sequence of the whole brain. Diffusion images are processed to generate isotopic apparent diffusion coefficient maps using dedicated software allowing for proper classification of the lesions. Transversal fluid-attenuated inversion recovery and transversal T2-weighted turbo spin-echo sequences are also performed. Slice thickness is 5mm for all sequences. Scans are read by an experienced neuroradiologist blinded to the clinical data. The presence, number, volume and location of all new focal diffusion abnormalities were recorded.

SECONDARY OUTCOMES:
Ipsilateral stroke (ischaemic stroke, intracerebral bleeding or both, with symptoms lasting more than 24 h) or death between treatment and 30 days after treatment | 30 days after treatment
  Stroke and transient ischaemic attack is defined according to the Valve Academic Research Consortium (VARC) recommendation. In case of stroke, the modified Rankin scale (mRS) is assessed to categorize the patient's level of functional independence during daily activities.

OTHER OUTCOMES:
Neurocognitive function postoperatively compared to preoperative status | at baseline before treatment and at 1-3 days after treatment, at discharge and at 3 months
  Examinations were performed at baseline, pre-discharge and 3 months thereafter. Neurological status is assessed by a detailed clinical examination protocol. Cognitive function is evaluated using three different standardized neuropsychological tests and the Mini-Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, West-German Heart Center Essen, University Duisburg-Essen, Essen, Germany

REFERENCES:
- [Derived] Wendt D, Kleinbongard P, Knipp S, Al-Rashid F, Gedik N, El Chilali K, Schweter S, Schlamann M, Kahlert P, Neuhauser M, Forsting M, Erbel R, Heusch G, Jakob H, Thielmann M. Intraaortic Protection From Embolization in Patients Undergoing Transaortic Transcatheter Aortic Valve Implantation. Ann Thorac Surg. 2015 Aug;100(2):686-91. doi: 10.1016/j.athoracsur.2015.03.119. PMID 26234838